CLINICAL TRIAL: NCT02100189
Title: Esophageal Cancer (10030139, 10066354) Screening With FISH in Esophageal Cytology
Brief Title: Esophageal Cytology With FISH in Detecting Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Hunter, Interim Dean, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00009213; NCI-2014-00384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00009213 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2014-02-28; First posted 2014-03-31 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia; Dysplasia; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Esophagitis; Gastroesophageal Reflux Disease; High Grade Dysplasia in Barrett Esophagus; Weight Loss
MeSH Terms: conditions — Deglutition Disorders; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Esophagitis; Gastroesophageal Reflux; Weight Loss | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening (esophageal cytology, FISH) (Experimental): Participants swallow the capsule (Oesotest from Actimed) and then wait 10 minutes before the sponge is pulled out through the esophagus by gentle traction on the string. Cytology samples from the sponge are harvested and analyzed by FISH. Participants then undergo standard EGD or upper endoscopy.
  Interventions: Other: Cytology Specimen Collection Procedure; Procedure: Esophagogastroduodenoscopy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo esophageal cytology collection
  Other Names: Cytologic Sampling
Procedure: Esophagogastroduodenoscopy — Undergo standard EGD or endoscopy
  Other Names: EGD
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies whether esophageal cytology plus fluorescence in situ hybridization (FISH) is equal to or better than esophago-gastro-duodenoscopy (EGD) or upper endoscopy for the early detection of esophageal cancer. Genes are the units of deoxyribonucleic acid (DNA) the chemical structure carrying genetic information that determine many human characteristics. Certain genes in cancer cells may determine how the tumor grows or spreads and how it may respond to different drugs. Part of this study is to test those genes in esophageal cells using FISH.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if sponge cytology with FISH is a reliable screening tool for esophageal dysplasia/cancer, and determine its sensitivity and specificity, compared to the gold standard procedure (upper endoscopy).

SECONDARY OBJECTIVES:

I. Determine if the cytology screening with FISH biomarkers is more cost effective than upper endoscopy for the screening of esophageal cancer and the surveillance of esophageal metaplasia and dysplasia.

II. Determine the limitations and future needs to improve this technique.

OUTLINE:

Participants swallow the capsule (Oesotest from Actimed) and then wait 10 minutes before the sponge is pulled out through the esophagus by gentle traction on the string. Cytology samples from the sponge are harvested and analyzed by FISH. Participants then undergo standard EGD or upper endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known esophageal cancer diagnosed by previous endoscopy

  * Adenocarcinoma
  * Squamous cell carcinoma
* Patients determined to be at risk for esophageal cancer:

  * Subjects with a history of Barrett's esophagus
  * Subjects with a history of low or high grade dysplasia
  * Subjects with a history of gastroesophageal reflux disease (GERD)
  * Subjects with a history of esophagitis
  * Subjects with symptoms of esophageal cancer (EC) referred for endoscopy (new onset dysphagia, weight loss, etc)
* Patients must be scheduled for a procedure capable of providing a definitive pathological diagnosis and evaluating for complications of the esophageal sponge on the same day as the study procedure, either:

  * Upper endoscopy
  * Surgical esophagectomy
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status =< 3 (Karnofsky >= 30%) will be included
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with severe, symptomatic dysphagia (unable to pass solids)
* Subjects that are unable to swallow a tablet/pill for any reason
* Subjects with a previous esophagectomy
* Subjects with esophageal varices
* Subjects unable to provide consent
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hunter, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Esophageal Cell Harvesting Procedure: Participants swallow the capsule (Oesotest from Actimed) and then wait 10 minutes before the sponge is pulled out through the esophagus by gentle traction on the string. Cytology samples from the sponge are harvested and analyzed by FISH. Participants then undergo standard EGD or upper endoscopy.
Period: Overall Study
Arm/Group | Esophageal Cell Harvesting Procedure
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Esophageal Cell Harvesting Procedure
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 50
Body Mass Index, average [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (7.66)
Number of participants with history of GERD [Count of Participants; unit: Participants] | 38
Number of participants with history of Barrett's Esophagus [Count of Participants; unit: Participants] | 28
Number of participants with a history of PPI use [Count of Participants; unit: Participants] | 39

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Sponge Cytology Using FISH
Description: All processed (FISH) esophageal cells will be compared to the final pathologic esophageal diagnoses determined by EGD or surgical resection to assess the test's sensitivity and specificity for the diagnosis of esophageal cancer. Using EGD diagnostic outcomes as the gold standard, the sensitivity and specificity will be computed with corresponding 95% confidence interval of the FISH sponge cytology test in the study population.
Time Frame: At the time of sponge cytology and EGD
Population: Analysis was per protocol
Measure: Number (95% Confidence Interval); unit: percentage of cases among positive tests
Arm/Group | Esophageal Cell Harvesting Procedure
Number analyzed (Participants) | 50
percentage of cases among positive tests | 13.3 [3.76 to 30.72]
Statistical Analysis 1: Comparison: Esophageal Cell Harvesting Procedure; Test type: Superiority or Other; Sensitivity; Sensitivity = 13.30, 95% CI 2-sided [3.76 to 30.72], Standard Error of Mean 0.062 — Exact Binomial confidence interval

2. Primary Outcome: Specificity of Sponge Cytology Using FISH
Description: as for outcome 1
Time Frame: At the time of sponge cytology and EGD
Population: Per protocol
Measure: Number (95% Confidence Interval); unit: Percentage of non-cases among neg tests
Arm/Group | Esophageal Cell Harvesting Procedure
Number analyzed (Participants) | 50
Percentage of non-cases among neg tests | 94.7 [73.97 to 99.87]
Statistical Analysis 1: Comparison: Esophageal Cell Harvesting Procedure; Test type: Superiority or Other; Specificity; Specificity = 94.7, 95% CI 2-sided [73.97 to 99.87], Standard Error of Mean 0.051 — Exact binomial confidence interval

3. Secondary Outcome: Adverse Events Associated With FISH Sponge Cytology Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Descriptive statistics will be used to summarize all adverse events associated with FISH sponge cytology test.
Time Frame: At the time of sponge cytology procedure
Population: Intent to Treat (ITT)
Measure: Number; unit: adverse events
Arm/Group | Esophageal Cell Harvesting Procedure
Number analyzed (Participants) | 50
adverse events | 16

4. Secondary Outcome: Tolerability of FISH Spongy Cytology
Description: Tolerability is defined as the patient's willingness to repeat procedure.
Time Frame: After completion of FISH and EGD
Population: Intent to Treat (ITT)
Measure: Number; unit: percentage of subjects tolerating test
Arm/Group | Esophageal Cell Harvesting Procedure
Number analyzed (Participants) | 50
percentage of subjects tolerating test | 100

ADVERSE EVENTS:
Time Frame: Adverse Events were collected on patients from time of consent to completion of cell harvesting procedure, up to 24 hours.
Arm/Group | Esophageal Cell Harvesting Procedure
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 16/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esophageal Cell Harvesting Procedure (N=50)
Gagging / Discomfort (Gastrointestinal disorders) | 14 (14) — Patients who either demonstrated gagging during the procedure and / or expressed discomfort immediately following the study procedure
Emesis (Gastrointestinal disorders) | 2 (2) — Patients who vomited during or immediately following study procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No